CLINICAL TRIAL: NCT01868282
Title: Comparison of Efficacy and Safety of Perihamstring Local Anesthetic Injection to Obturator Nerve Block When Combined With Subsartorial Saphenous Block for Anterior Cruciate Ligament Repair. A Randomized Double Blinded Study.
Brief Title: Study of Pain Management Techniques Following Anterior Cruciate Ligament Repair Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103681
Record Dates: First submitted 2013-04-26; First posted 2013-06-04 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: anterior cruciate ligament repair, Obturator nerve block, Hamstrings graft, Ropivacaine,; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Hamstrings block
  Interventions: Procedure: Hamstrings block
- Group 2 (Active Comparator): Obturator block
  Interventions: Procedure: Obturator block
- Group 3 (Sham Comparator): Control group
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Hamstrings block — patients enrolled in the study will receive subsartorial saphenous nerve block in all the three groups. Patients in group 1 will receive perimuscular injections around the gracilis and semi-tendinosus muscles. The needle is redirected to the fascial plane between Sartorius and gracilis muscle after the sub-sartorial canal block where 7.5 ml of 0.5% ropivacaine is injected around the muscle. The needle is further advanced to the fascial planes between semimembranosus and semitendinosus and an additional 7.5 ml of 0.5% ropivacaine will be injected around the semitendinosus muscle. Following this a sham injection of 10mL of saline for the anterior division of obturator nerve will also be performed as in group 2 to ensure blinding.
  Other Names: perimuscular injections
  Arms: Group 1
Procedure: Obturator block — Patients in group 2 will receive anterior division of obturator nerve block along with subsartorial canal block. After ensuring aseptic precautions, the saphenous nerve block is performed similar to that as in group 1. The anterior branch of obturator nerve will be visualised in the proximal thigh medial to femoral vessels between adductor longus and adductor brevis. A 22 gauge 90 mm PNS block needle will be inserted under ultrasound guidance to reach the anterior division of obturator nerve confirmed with neurostimulation followed by injection of 10 ml of 0.5% ropivacaine around the nerve. This group will receive sham injection of 15mL of saline around semitendinosus and semimembranosus as in group 1
  Other Names: anterior division obturator nerve block
  Arms: Group 2
Procedure: Control group — The patients in group 3 will form the control group. After performance of the subsartorial saphenous nerve block, patients in group 3 will receive sham injections of saline for the obturator nerve block and the hamstrings block (perimuscular injections).
  Other Names: saline group
  Arms: Group 3

SUMMARY:
Patients scheduled to undergo knee arthroscopy with anterior cruciate ligament repair with graft from the ipsilateral hamstrings and gracilis will be randomized to one of three groups. All patients will receive subsartorial saphenous nerve block. Along with this, Group 1 will receive perihamstring local anesthetic infiltration (Hamstring block), Group 2 will receive blockade of the anterior division of obturator nerve and Group 3 (control group) will receive sham injections of hamstrings and anterior division obturator nerve. All patients will receive co-analgesics for home discharge. The study will evaluate the efficacy of subsartorial saphenous nerve block alone or in combination with either hamstring block or obturator block with regards to postoperative analgesia especially the donor site pain and total analgesic consumption.

DETAILED DESCRIPTION:
Performance of arthroscopic knee repairs on day care basis necessitates adequate post-operative analgesia for successful home discharge since post-operative pain is known to be the commonest cause of unanticipated readmissions of day care patients. Early return to activity is also crucial to ensure adequate surgical outcomes. Anterior cruciate ligament (ACL) repair is commonly performed by arthroscopic approach with an ipsilateral hamstring-gracilis graft. This has shown to be superior to patellar tendon grafts with regards to pain and functional outcomes after surgery. Postoperative pain from the graft donor site and anterior knee pain form the surgery can lead to decreased range of motion and poor rehabilitation. A variety of regional anesthetic techniques are being tried for out-patient knee surgery like spinal adjuvants; intra and peri-articular injection, single injection and continuous blocks of the femoral and sciatic nerves, oral pills and cryoanalgesia. Opioid based analgesia with or without co-analgesics is not suited for dynamic pain relief since Aα and Aδ nerve fibres that carry pain are poorly inhibited by opioids while effectively inhibited by local anesthetics. Multimodal analgesic regimens work well for ambulatory surgeries especially when combined with regional analgesic techniques. Regional techniques decrease opioid consumption and hence opioid related side effects. Intra and peri-articular injections have a short duration of action compared to nerve blocks apart from the concerns of chondrotoxicity of intra-articular local anesthetics. Although femoral- and sciatic nerve blocks provide adequate analgesia, the weakness of the quadriceps and hamstrings can prevent early rehabilitative efforts and also pose a risk for patient falls following home discharge. Hence, novel regional techniques of analgesia like blocking the infrapatellar branch of saphenous nerve, graft site injections of local anesthetics through the arthroscopic sleeve and single injection adductor canal block have been tried. Isolated sensory block of the surgical and graft site without motor block is the Holy Grail in search for these ambulatory patients.

Saphenous nerve, the terminal branch of femoral nerve supplies the majority of the knee joint. The femoral nerve exits the adductor canal and gives the terminal branch of saphenous nerve which lies between the Sartorius muscle and femoral artery in the sub-sartorial canal. Subsartorial canal block has been successfully utilized for forefoot surgery and knee arthroplasty but this has not been evaluated for ACL repairs. Saphenous nerve can be successfully blocked in the subsartorial canal without the risks of leg weakness but this alone is insufficient to provide analgesia to the graft donor site which is usually the gracilis tendon and the hamstrings tendon. Depositions of local anesthetics around the harvested muscle or blockade of the nerve supplying it are attractive strategies to decrease donor site pain but have not been explored for this purpose in a randomized fashion. The investigators hypothesize that the combination of any of the above two techniques to decrease donor site pain along with subsartorial saphenous nerve block can provide adequate analgesia in these patients. The anterior branch of the obturator nerve needs to be blocked since it supplies the gracilis muscle. To decrease the donor site pain, the saphenous nerve block can be combined with block of the anterior branch of obturator nerve. Alternatively, the saphenous nerve block can be combined with deposition of local anesthetic around the graft donor muscles. The extent to which the two techniques benefit the patients in terms of overall analgesia and the graft site analgesia has not been evaluated. With this background, the investigators want to compare the analgesic efficacy of subsartorial saphenous nerve block with either perihamstrings infiltration or blockade of the anterior division of obturator nerve in patients undergoing ACL reconstruction with ipsilateral autograft from gracilis and hamstring muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of 16-85years of age, scheduled to undergo anterior cruciate ligament repair with ipsilateral hamstrings graft.
2. ASA Class I-III

Exclusion Criteria:

1. ASA 4
2. Revision surgery
3. Graft harvest from the contralateral hamstrings or allograft
4. Narcotic dependent (opioid intake more than 3 months) or any chronic pain conditions
5. Patients with associated significant cardiac and respiratory disease
6. Patients with coexisting hematological disorder or with deranged coagulation parameters.
7. Patients with pre-existing major organ dysfunction such as hepatic and renal failure.
8. Psychiatric illnesses
9. Emergency surgery
10. Lack of informed consent.
11. Allergy to any of the drugs used in the study
12. Preoperative neurological deficits

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Post-operative pain scores at admission to PACU | Baseline
  The primary outcome will be post-operative pain scores at I hour after arrival in PACU.

SECONDARY OUTCOMES:
Pain scores at 4 hours of arrival to PACU | 4 hours
  patients will be assessed for pain scores at rest and movement after 4 hours of arrival to the recovery from the operating room

OTHER OUTCOMES:
first 24 pain scores | Day1
  Patients will be provided with a diary to document pain scores every 6 hourly thereafter until 24 hours after their time of arrival in PACU (time 0). Patients will be discharged home along with a data collection sheet for documenting pain scores, analgesic consumption and side effects at various time intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Sugantha Ganapathy, FRCPC, Principal Investigator — London Health sciences Center, Western University, London, Ontario, Canada; N6A5A5
Locations (1):
- University Hospital, London Health Sciences Center,, London, Ontario, Canada

REFERENCES:
- [Background] Bushnell BD, Sakryd G, Noonan TJ. Hamstring donor-site block: evaluation of pain control after anterior cruciate ligament reconstruction. Arthroscopy. 2010 Jul;26(7):894-900. doi: 10.1016/j.arthro.2009.11.022. Epub 2010 May 13. PMID 20620788
- [Background] Saranteas T, Anagnostis G, Paraskeuopoulos T, Koulalis D, Kokkalis Z, Nakou M, Anagnostopoulou S, Kostopanagiotou G. Anatomy and clinical implications of the ultrasound-guided subsartorial saphenous nerve block. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):399-402. doi: 10.1097/AAP.0b013e318220f172. PMID 21697687
- [Background] Lundblad M, Forssblad M, Eksborg S, Lonnqvist PA. Ultrasound-guided infrapatellar nerve block for anterior cruciate ligament repair: a prospective, randomised, double-blind, placebo-controlled clinical trial. Eur J Anaesthesiol. 2011 Jul;28(7):511-8. doi: 10.1097/EJA.0b013e32834515ba. PMID 21455076
- [Background] Buckenmaier CC 3rd. Anaesthesia for outpatient knee surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):255-70. doi: 10.1053/bean.2002.0237. PMID 12491556
- [Derived] Johnston DF, Sondekoppam RV, Uppal V, Litchfield R, Giffin R, Ganapathy S. Effect of combining peri-hamstring injection or anterior obturator nerve block on the analgesic efficacy of adductor canal block for anterior cruciate ligament reconstruction: a randomised controlled trial. Br J Anaesth. 2020 Mar;124(3):299-307. doi: 10.1016/j.bja.2019.11.032. Epub 2020 Jan 21. PMID 31980156